CLINICAL TRIAL: NCT03715023
Title: A Double Blind, Placebo-controlled Study to Assess the Anti-viral Effect, Safety and Tolerability of Inhaled PC786 for the Treatment of Acute Respiratory Syncytial Virus (RSV) Infection in Adult Hematopoietic Stem Cell Transplant Recipients
Brief Title: Anti-viral Effect of PC786 on RSV Infection on HSCT Recipients
Acronym: TreatRSV1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Practical issues that could not be resolved resulting in recruitment difficulties at sites.
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC_RSV_004; 2018-001667-24 (EudraCT Number)
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV infection; Hematopoeitic stem cell transplant
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — PC-786

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active + SoC (Experimental): Daily doses of PC786 for 3 days + SoC
  Interventions: Drug: PC786; Drug: SOC
- Placebo + SoC (Placebo Comparator): Daily doses of Placebo for 3 days + SoC
  Interventions: Drug: Placebo; Drug: SOC

INTERVENTIONS:
Drug: PC786 — PC786 suspension for inhalation
  Arms: Active + SoC
Drug: Placebo — Placebo solution for inhalation
  Arms: Placebo + SoC
Drug: SOC — Standard treatment for RSV infection at study site

SUMMARY:
This study tests the effects of an experimental drug PC786 in people infected with Respiratory Syncytial Virus (RSV). PC786 may be useful in treating patients infected with RSV as it works by interfering with the way the virus multiplies. PC786 is an inhaled medicine. Participants will be treated with SoC treatment (e.g. oral ribavirin and/or IV immunoglobulin), half of the participants will receive PC786 in addition and half will receive a placebo treatment. The study will take place at multiple sites in UK and will include approximately 30 participants. The maximum study duration will be about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Received an allogeneic or autologous hematopoietic stem cell transplant (HSCT) using any conditioning regimen
* Experienced new onset of at least one of the following respiratory symptoms ≤5 days before study Day 1:

Nasal congestion or stuffiness, runny nose (rhinorrhoea), cough, or sore throat OR Worsening of at least one of those symptoms, if symptoms are chronic OR Wheezing, sputum production, pleuritic chest pain, increased respiratory rate, signs on chest auscultation, hypoxia, increased supplemental oxygen requirement or new infiltrates on chest X-ray/CT

* A positive RSV diagnostic test
* Provided written informed consent

Exclusion Criteria:

* Is intubated and requires invasive ventilation
* Has received any investigational RSV vaccine after HSCT, or has received any monoclonal anti-RSV antibodies within 4 months or 5 half-lives before participation
* Treatment with intravenous ribavirin
* Positive for test for influenza or parainfluenza
* Significant untreated bacteraemia or fungaemia
* Significant untreated bacterial, fungal, or viral pneumonia
* Precluded from participating as a result of treatment with another investigational drug or participation in another clinical trial
* Other disease or condition which would preclude the subject's participation in a clinical trial
* Is receiving an antiretroviral protease inhibitor
* Has chronic, active hepatitis infection
* Known alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
RSV viral load measured in nasal secretions by reverse transcription quantitative PCR (RT-qPCR) | Day 1 to Day 3
Proportion of participants reporting one or more treatment-emergent adverse event (TEAE) | Baseline to Day 28
Proportion of participants who discontinue due to an adverse event | Baseline to Day 28
Proportion of participants who meet the markedly abnormal criteria for 12-lead ECG assessment at lease once post dose | Baseline to Day 28
Proportion of participants who meet the markedly abnormal criteria for vital signs assessment at lease once post dose | Baseline to Day 28
Proportion of participants who meet the markedly abnormal criteria for safety laboratory assessment at lease once post dose | Day 1 to Day 28
Proportion of participants who meet the markedly abnormal criteria for peak expiratory flow assessment at lease once post dose | Day 1 to Day 28

SECONDARY OUTCOMES:
Average change in RSV load measured in nasal secretion | Day 1 to Day 7
Change in RSV load in nasal secretion | Baseline to Day 3
Change in RSV load in nasal secretion | Baseline to Day 7
Duration in viral shedding measured in nasal secretion | Day 1 to Day 28
Determination of nasal concentrations of PC786 | Days 1, 2, 3, 7, 14 and 28
Maximum observed concentration (Cmax) of PC786 measured in plasma | Day 1, Pre-dose to 4 hours
Trough plasma concentration (Ctrough) of PC786 | Days 2 and 3, Pre-dose
Area under the concentration versus time curve from time zero to time at 4 hours (AUC0-4) of PC786 in plasma | Day 1, Pre-dose to 4 hours
Last quantifiable concentration (Ct last) of PC786 measured in plasma | Day 1, and multiple timepoints to Day 28
Changes in RSV symptoms measured using a symptom diary card | Days 1, 2, 3, 4, 5, 6, 7, 14 and 28
Proportion of participants developing lower respiratory tract infection (LRTI) or pneumonia | Day 1 to 28
Proportion of participants progressing to invasive ventilation | Day 1 to 28
Trends in oxygen saturation index | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Alison Murray, Study Director — Pulmocide Ltd
Locations (7):
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - St Georges University Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield